CLINICAL TRIAL: NCT03791905
Title: A Phase II Randomized Trial of PET Imaging in Assessing Response to Induction Chemotherapy in Esophageal Squamous Cell Carcinoma Treated With Definitive Chemoradiotherapy
Brief Title: PET Imaging-guided Chemoradiotherapy in Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mian XI (Other)
Responsible Party: Sponsor-Investigator, Mian XI, Associate Preofessor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PETESCC
Record Dates: First submitted 2018-12-31; First posted 2019-01-03 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Neoplasm, Esophageal; Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; PET; Definitive chemoradiotherapy; Induction chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell; Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Cisplatin; Oxaliplatin; Fluorouracil; Leucovorin; Radiotherapy, Intensity-Modulated; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: Randomized parallel study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TP Arm (Experimental): Patients with baseline PET scan assigned to this Arm will receive two cycles of 3-weekly schedule of induction chemotherapy with paclitaxel/cisplatin (TP), consisting of paclitaxel 150 mg/m2 on day 1 and cisplatin 75 mg/m2 on day 1. Repeat PET was performed on days 36-42 and changes in SUVmax from baseline were assessed. PET responders (≥35% decrease in SUVmax) continued on the same chemotherapy regimen during radiotherapy, whereas PET non-responders (<35% decrease in SUVmax) crossed over to FOLFOX regimen concomitantly with radiation. All patients received external-beam radiation using intensity-modulated radiotherapy. The prescribed dose is generally 50-60 Gy in 25-28 fractions.
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy; Device: PET
- FOLFOX Arm (Experimental): Patients with baseline PET scan assigned to this Arm will receive three cycles of 2-weekly schedule of induction chemotherapy with FOLFOX (oxaliplatin, leucovorin, 5-FU), consisting of oxaliplatin 85 mg/m2 on day 1, leucovorin 400 mg/m2, and 5-FU 2 g/m2 on day 1. Repeat PET was performed on days 36-42 and changes in SUVmax from baseline were assessed. PET responders (≥35% decrease in SUVmax) continued on the same chemotherapy regimen during radiotherapy, whereas PET non-responders (<35% decrease in SUVmax) crossed over to TP regimen concomitantly with radiation. All patients received external-beam radiation using intensity-modulated radiotherapy. The prescribed dose is generally 50-60 Gy in 25-28 fractions.
  Interventions: Drug: Oxaliplatin; Drug: 5-FU; Drug: Leucovorin; Radiation: Intensity-modulated radiotherapy; Device: PET

INTERVENTIONS:
Drug: Paclitaxel — chemotherapy drug
  Other Names: Taxol
  Arms: TP Arm
Drug: Cisplatin — chemotherapy drug
  Other Names: DDP
  Arms: TP Arm
Drug: Oxaliplatin — chemotherapy drug
  Other Names: OXA
  Arms: FOLFOX Arm
Drug: 5-FU — chemotherapy drug
  Other Names: Fluorouracil
  Arms: FOLFOX Arm
Drug: Leucovorin — chemotherapy drug
  Other Names: CF
  Arms: FOLFOX Arm
Radiation: Intensity-modulated radiotherapy — radiotherapy technique
  Other Names: IMRT
Device: PET — Using PET to evaluate response to induction chemotherapy
  Other Names: PET-CT

SUMMARY:
Since multiple studies have demonstrated that PET can identify responders and non-responders to induction chemotherapy, using FDG-PET imaging to guide treatment decisions has prompted interest in clinical practice. The aim of this study was to evaluate whether changing chemotherapy regimen during radiation based on PET response to induction chemotherapy can improve clinical complete response (cCR) in patients with unresectable esophageal squamous cell carcinoma (ESCC).

DETAILED DESCRIPTION:
A total of 216 patients with baseline PET scan were randomized to one of 2 induction chemotherapy arms: paclitaxel/cisplatin (TP) on days 1, 22 or FOLFOX (oxaliplatin, leucovorin, 5-FU) on days 1, 15, 29. Repeat PET was performed on days 36-42 and changes in max standardized uptake value (SUVmax) from baseline were assessed. Using a predefined cut-off value of a 35% decrease in SUVmax, PET responders (≥35% decrease in SUVmax) continued on the same chemotherapy regimen during radiotherapy, whereas PET non-responders (<35% decrease in SUVmax) crossed over to an alternative chemotherapy regimen concomitantly with radiation. All patients received external-beam radiation using intensity-modulated radiotherapy. The prescribed dose is generally 50-60 Gy in 25-28 fractions, 5 days per week.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the esophagus;
2. Absence of hematogenous metastasis disease, confirmed by endoscopic ultrasound (EUS) and PET-CT scan (according to UICC TNM version 8);
3. Not suitable for surgery (either for medical reasons or patient's choice);
4. Age at diagnosis 18 to 70 years;
5. Eastern Cooperative Oncology Group performance status ≤ 2
6. No prior cancer therapy;
7. No history of concomitant or previous malignancy;
8. Hematologic function: WBC ≥ 4.0×109/L, PLT ≥ 80×109/L, Hb ≥ 10mg/dL;
9. Renal function: Cr ≤ 1.25×UNL;
10. Hepatic function: BIL ≤ 1.5×UNL, ALT/AST ≤ 2.5×UNL;
11. Documented informed consent to participate in the trial.

Exclusion Criteria:

1. Younger than 18 or older than 70 years of age;
2. ECOG performance status of 3 or above;
3. Other cancer history;
4. Previous radiotherapy history;
5. Subjects with distant metastases;
6. Pregnancy or breast feeding. Women of childbearing age must use effective contraception;
7. Serious cardiovascular disease (congestive heart failure, uncontrollable arrhythmia, unstable angina, myocardial infarction, serious heart valve disease, resistant hypertension);
8. Evidence of bleeding diathesis or serious infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
clinical complete response | 3 months after the treatment (plus or minus 7 days)
  RECIST (Response Evaluation Criteria in Solid Tumors) criteria was used to determine the tumor response. Tumor response was evaluated 3 months after the completion of treatment based on CT or PET-CT scans, endoscopy with biopsies.

SECONDARY OUTCOMES:
Overall survival | 3 years after randomization
  From the enrollment to the date of death from any cause or date of lost follow-up
Progression-free survival | 3 years after randomization
  From the date of randomization to the date of disease progression or last follow-up
Chemoradiotherapy-related toxicity | From the date of randomization to the 3 months after treatment
  Treatment-related toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Mian XI, MD, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ku GY, Kriplani A, Janjigian YY, Kelsen DP, Rusch VW, Bains M, Chou J, Capanu M, Wu AJ, Goodman KA, Ilson DH. Change in chemotherapy during concurrent radiation followed by surgery after a suboptimal positron emission tomography response to induction chemotherapy improves outcomes for locally advanced esophageal adenocarcinoma. Cancer. 2016 Jul 1;122(13):2083-90. doi: 10.1002/cncr.30028. Epub 2016 May 6. PMID 27152857